CLINICAL TRIAL: NCT07287345
Title: Adjunctive Colchicine's Effect on Inflammatory Markers and Corresponding New-Onset Atrial Fibrillation Rates Post Coronary Artery Bypass Graft Procedure: A Pilot Study
Brief Title: Colchicine's Effect on Inflammatory Markers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ayesha Ather (Other)
Responsible Party: Sponsor-Investigator, Ayesha Ather, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102331
Record Dates: First submitted 2025-12-01; First posted 2025-12-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Colchicine; Inflammation in Cardiac Surgery; Post Operative Atrial Fibrillation; Inflammatory Markers; Colchicine Adverse Reaction
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care and placebo (Placebo Comparator): placebo capsule
  Interventions: Drug: Placebo
- Standard of care and colchicine (Experimental): colchicine capsule
  Interventions: Drug: Colchicine (Colcrys®)

INTERVENTIONS:
Drug: Colchicine (Colcrys®) — Colchicine dosing is based on actual body weight and renal function (creatinine clearance). Subjects will initiate study medication (placebo or active drug) 5 days prior to surgery and continue therapy for 10 days postoperatively or until hospital discharge, whichever occurs first.
  For patients weighing ≥70 kg:
  If CrCl >30 mL/min: Colchicine 0.6 mg twice daily
  If CrCl <30 mL/min: Colchicine 0.3 mg once daily
  For patients weighing <70 kg:
  If CrCl >30 mL/min: Colchicine 0.6 mg once daily
  If CrCl <30 mL/min: Colchicine 0.3 mg every other day
  Arms: Standard of care and colchicine
Drug: Placebo — Placebo dosing is based on actual body weight and renal function (creatinine clearance). Subjects will initiate study medication (placebo or active drug) 5 days prior to surgery and continue therapy for 10 days postoperatively or until hospital discharge, whichever occurs first.
  For patients weighing ≥70 kg:
  If CrCl >30 mL/min: Placebo 0.6 mg twice daily
  If CrCl <30 mL/min: Placebo 0.3 mg once daily
  For patients weighing <70 kg:
  If CrCl >30 mL/min: Placebo 0.6 mg once daily
  If CrCl <30 mL/min: Placebo 0.3 mg every other day
  Arms: Standard of care and placebo

SUMMARY:
This study wants to see if the medicine colchicine can help lower inflammation and reduce the chance of developing an irregular heartbeat (atrial fibrillation) after heart bypass surgery. Adults having coronary artery bypass surgery (CABG) can join. Participants will be randomly placed into one of two groups: one group will receive colchicine along with usual care, and the other will receive a placebo (a look-alike capsule with no medicine) along with usual care. Everyone will take a study capsule, and neither the patients nor the study team will know which capsule is being given. Everyone in the study will take study capsule, and neither the patients nor the study team will know who is receiving colchicine or placebo. Blood samples and health information will be collected before surgery; at 24, 48, 72, and 96 hours after surgery; and again at 10 days after surgery or at hospital discharge, whichever comes first. The investigators will look at inflammation marker levels, whether atrial fibrillation happens, and any side effects. This small study will help to generate effect size estimates and safety data that will help plan a larger study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Coronary artery bypass graft (CABG) planned procedure

Exclusion Criteria:

* History of atrial fibrillation
* Off-pump CABG procedure
* Current treatment with colchicine for any cause
* Hypersensitivity to colchicine (as indicated by rash; hives; itching; red, swollen, blistered, or peeling skin with or without fever)
* Emergency cardiac surgery
* Extracorporeal Membrane Oxygenation (ECMO) pre- or post-cardiac surgery
* Heart transplant patients
* Left ventricular assist device (LVAD) patients
* Serum creatinine >2.0 mg/dL
* Preoperative elevated CK or known myopathy
* Severe liver disease or elevation of serum transaminases (>1.5 times the upper limit of 40 units/liter)
* Chronic intestinal disease or blood dyscrasia
* Unable to speak English
* Pregnancy or lactation in women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory markers | Baseline (pre-surgery), 24, 48, 72, 96 hours post-surgery and 10 days postoperatively or at discharge, whichever occurs first.
  markers of inflammation (IL-6, CRP, IL-18, IL-1β, IL-8, and TNF-α) will be measured at predefined time points. Blood samples will be obtained as part of routine clinical care and analyzed using commercially available ELISA assays.
Rate of post-operative atrial fibrillation (POAF) | Through discharge (up to 15 days)
  Postoperative atrial fibrillation (POAF) incidence will be assessed through daily chart review.

SECONDARY OUTCOMES:
Number of participants discontinuing treatment | Through discharge (up to 15 days)
  treatment discontinuation rates due to adverse events will be measured
Change in Liver Function | Baseline and Post operatively (approximately 24 hours)
  Assessed as the impact on clinical biomarkers, i.e., ALT, AST in units per liter.
Change in creatinine level | Baseline through discharge (up to 15 days)
  Assessed as the impact on clinical biomarkers, i.e., creatinine level in mg/dl
Creatine kinase level | Through discharge (up to 15 days)
  Assessed as the impact on clinical biomarkers, creatine kinase (i.e., CK level) in units per liter
Complete blood count (CBC). | Through discharge (up to 15 days)
  Assessed as the impact on clinical biomarker complete blood count (CBC).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sekela, MD, Study Director — University of Kentucky
Locations (1):
- University of Kentucy, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No